CLINICAL TRIAL: NCT03731962
Title: Using Preprocedural Urine NMR-Based Metabolomics Analysis to Prediction the Risk of Contrast Induced Nephropathy Following Elective Coronary Angiography
Brief Title: Using Preprocedural Urine NMR(Nuclear Magnetic Resonance) -Based Metabolomics Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SBMU23567/J
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Contrast-induced Nephropathy; Coronary Angiography
Keywords: Urine Metabolomics; Contrast Induced Nephropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Developed Contrast Induced Nephropathy (Active Comparator): Coronary Angiography
  Interventions: Procedure: Coronary Angiography
- Without CIN (Other): Coronary Angiography
  Interventions: Procedure: Coronary Angiography

INTERVENTIONS:
Procedure: Coronary Angiography — All patients received approximately 60 mL of intra arterial iodinated contrast material that was administered via computer-controlled automated power injector at 4 mL per second.

SUMMARY:
The use of coronary intervention has increased over the last decade. Contrast induced nephropathy (CIN) that develops as a result of procedures using intravenous or intra arterial contrast enhancement, or other diagnostic procedures, has been reported to be the third leading cause of acute renal failure in hospitalized patients. It has been hypothesized that this occurs as a result of direct toxicity, oxidative stress, and ischemic injury. Numerous studies have evaluated the incidence of CIN in patients undergoing angiography. There are limited studies in the acute care setting. Therefore, a tool that could identify early risk factors for CIN would be valuable for patient care.

Metabolomic profiling is the identification of small molecule metabolites that are altered in response to injury. We hypothetize that urine metabolomic profiles may differ in patients before and after contrast administration coronary intervention.We hypothesized that metabolomic profiles will differ between those patients who develop CIN and those who do not after contrast administration. In addition we believe that metabolomics profiles prior to angiography may identify subjects who will go on to develop CIN and are therefore at higher risk.

DETAILED DESCRIPTION:
The specific aim of this pilot study is to determine if metabolomics profiles differ in patients who develop CIN after contrast administration for coronary angiography versus those who do not. Additionally, our goal was to identify specific urinary metabolites that warrant further investigation.This is a pilot study of prospectively identified patients undergoing a coronary intervention with intraarterial contrast during their evaluation. The study was approved by the University of Shahid Beheshti, Medical institutional review boards.

100 number of patients were enrolled. To be eligible for the study, patients had to be >18 years old, undergoing coronary angiography and have at least 1 of the following high risk features for CIN: diabetes, coronary artery disease, congestive heart failure. Past medical history was confirmed by chart review if available, or patient report.

Patients were excluded from the study if they had an estimated glomerular filtration rate <15 mL/min/1.73 m2, a history of organ transplantation, were currently on immunosuppressive medications, were septic or on antibiotic therapy, had a history of or were currently receiving dialysis of any type, had an exposure to iodinated contrast within 3 days prior to the study, or had multiple doses of contrast given.

Patients were managed according to the treating provider recommendations. No intervention was requested as part of this study. There was no institutional standard for mandatory fluid administration or use of N-acetylcysteine prior to elective coronary angiography.All patients received approximately 60 mili Liter of intravenous iodinated contrast material that was administered via computer-controlled automated power injector at 4 mL per second.

data were collected prospectively after patients were identified as fulfilling inclusion and exclusion criteria, and informed consent was obtained. Data collection included , demographics, dietary history, medical history, physical examination, and electrocardiogram findings, as documented by the treating emergency physician. Medical history was confirmed through patient self-report and review of the medical record when available. Medications administered before arrival were also recorded. No additional laboratory tests were mandated as a part of the trial study and the treating physician ordered all tests, except urinary metabolomics analysis, according to their clinical judgment. Urine samples were collected as a midstream sample or via a foley bag prior to angiography and 12 hours post imaging. Samples were aliquoted into 2 mL samples and frozen at -80˚C.

Serum creatinine levels were recorded at presentation, and at 24 and 72 hours. The outcome measure was the presence CIN, which was defined as an increase in serum creatinine level of ≥0.5 mg/dL above baseline within 72 hours after contrast administration.

ELIGIBILITY:
Inclusion Criteria:

* patients had to be >18 years old Undergoing elective coronary angiography

Exclusion Criteria:

* estimated glomerular filtration rate <15 mL/min/1.73 m2
* history of organ transplantation
* using immunosuppressive medications
* septic patients or on antibiotic therapy
* a history of receiving dialysis of any type
* an exposure to iodinated contrast within 3 days prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
developing CIN | within 48 hours after contrast administration
  an increase in serum creatinine level of ≥0.5 mg/dL above baseline within 48 hours after contrast administration

SECONDARY OUTCOMES:
Urine Metabolomics | within 48 hours after contrast administration
  Finding differences between urine metabolites profile between patients develop CIN and without CIN

CONTACTS AND LOCATIONS:
Overall Officials: Dalili, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Nooshin Dalili, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No